CLINICAL TRIAL: NCT05657587
Title: A Post Market Observational Case Series Study of Percutaneous Peripheral Nerve Stimulation (PNS) for the Treatment of Chronic Shoulder Pain
Brief Title: Treatment of Shoulder Osteoarthritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gramercy Pain Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0001
Record Dates: First submitted 2022-08-10; First posted 2022-12-20 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Chronic Shoulder Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- PNS Group: All subjects will receive the PNS device. The Sprint system delivers mild electrical stimulation to the shoulder. The Sprint system includes up to two leads (small wires) that are placed through your skin in your shoulder. The leads attach to devices worn on your body that delivers stimulation (stimulators).
  Interventions: Device: SPRINT PNS

INTERVENTIONS:
Device: SPRINT PNS — Each subject will have 2 leads placed for 60 days. The Sprint system delivers mild electrical stimulation to the shoulder. The Sprint system includes up to two leads (small wires) that are placed through your skin in your shoulder. The leads attach to devices worn on your body that delivers stimulation (stimulators).

SUMMARY:
The purpose of this study is to learn if pain can be relieved by delivering small amounts of electricity ("electrical stimulation") to the nerves relaying sensory information to the shoulder. This study will use a device called Sprint PNS system. PNS stands for Peripheral Nerve Stimulation. This device is cleared by the FDA for up to 60 days of use for relief of chronic or acute pain.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosed with degenerative changes within the shoulder complex

Key Exclusion Criteria:

* Pain exclusively in the anterior aspect of the shoulder
* Opioids for any condition other than shoulder pain
* Other implanted electronic device

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pain due to degenerative changes in the shoulder scheduled for commercial placement of the Sprint PNS system
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Reduction in average pain and/or reduction in pain interference | 15 days, 1 month, 2 months, 3 months, 6 months, and 12 months post Start of Treatment
  Average pain intensity is measured using the PROMIS-29 v2.0 profile. The measure assesses pain intensity using a single 0-10 numeric rating scale. Average pain interference is measured using Brief Pain Inventory--Short Form Question #9 (BPI-9). BPI-9 uses a 0-10 numeric rating scale across seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance.)

SECONDARY OUTCOMES:
Changes in pain intensity | baseline, start of treatment (lead placement); 15 days, 1 month, 2 months, 3 months, 6 months, and 12 months post Start of Treatment
  Changes in pain intensity will be assessed using the PROMIS-29 v2.0 profile. The measure assesses pain intensity using a single 0-10 numeric rating scale.
Changes in pain interference | baseline, start of treatment (lead placement); 15 days, 1 month, 2 months, 3 months, 6 months, and 12 months post Start of Treatment
  Changes in average pain interference are measured using Brief Pain Inventory--Short Form Question #9. The measure assesses pain interference using a 0-10 numeric rating scale across seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance.)
Range of motion of the shoulder | baseline, start of treatment (lead placement); 2 months, 3 months, 6 months, and 12 months post Start of Treatment
  Shoulder range of motion is measured as degrees of active range of motion based on physical examination.
Changes in Shoulder Function | baseline, start of treatment (lead placement); 15 days, 1 month, 2 months, 3 months, 6 months, and 12 months post Start of Treatment
  Shoulder function is measured using the Western Ontario Arthritis of the Shoulder (WOOS) index. The WOOS index is a patient-reported, disease-specific questionnaire for the measurement of the quality-of-life in patients with osteoarthritis.

CONTACTS AND LOCATIONS:
Locations (1):
- Gramercy Pain Center, Holmdel, New Jersey, United States